CLINICAL TRIAL: NCT06798090
Title: Evaluation of Clinical Success and Changes in Periodontal Tissues of Band-Loop Space Maintainers Produced With Three-Dimensional Printer and Conventional Technique
Brief Title: Evaluation of Band-Loop Space Maintainers Produced With Three-Dimensional Printer and Conventional Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sultan KELES, Associate Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/21
Record Dates: First submitted 2024-10-06; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Dental Health; Space Maintainer; Pediatric Dentistry; 3D Printing
Keywords: three dimensional printer; band and loop space maintainer; digital dentistry; PLAP-1; TNF-a
MeSH Terms: interventions — Chromosome Banding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Band and Loop Space Maintainer Produced with Three-Dimensional Printer (Study Group) (Experimental): Digital impressions will be taken with 3Shape intraoral scanner. Space maintainer will be designed with CAD/CAM technology. The three-dimensional printer to be used is HBD - 150D Dual Laser, and production will be made by micro laser sinterisation method from nickel - chromium weighted metal powders.
  Interventions: Device: Band and Loop Space Maintainer Produced with Three-Dimensional Printer
- Band and Loop Space Maintainer Produced with Conventional Technique (Control Group) (Active Comparator): For conventional production, impressions will be taken with traditional impression spoons using alginate material. Stainless steel appropriate band will be chosen according to the size of the abutment teeth, then will be send to the laboratory for soldering.
  Interventions: Device: Band and Loop Space Maintainer Produced with Conventional Technique

INTERVENTIONS:
Device: Band and Loop Space Maintainer Produced with Three-Dimensional Printer — Band and loop space maintainer produced with three-dimensional printer using micro laser sinterisation method
  Arms: Band and Loop Space Maintainer Produced with Three-Dimensional Printer (Study Group)
Device: Band and Loop Space Maintainer Produced with Conventional Technique — Band and loop space maintainer produced with conventional methods
  Arms: Band and Loop Space Maintainer Produced with Conventional Technique (Control Group)

SUMMARY:
Our research is planned as a randomised clinical trial. The main aim of our study is to evaluate the clinical success of band and loop space maintainers produced by three-dimensional printer and conventional technique and the changes they cause in periodontal tissues.

DETAILED DESCRIPTION:
Participants will be selected by simple random selection from systemically healthy children who will need bilateral lower deciduous first molar extraction and space maintainer application from patients who apply to Aydın Adnan Menderes University Faculty of Dentistry, Department of Pedodontics for treatment.

The study will be carried out in a split-mouth design, and it is planned to place a band and loop space maintainer produced by conventional technique on one side and a band and loop space maintainer produced with a three-dimensional printer on the other side in the lower jaw. The clinical success of these two appliances and the changes in periodontal tissues will be compared. In order to evaluate the clinical success, the survival of the appliances and the determined failure criteria (Dissolution of the bonding cement, Separation/breakage from solder area, Embedding of the space maintainer inside towards the gum, Loop distortion/breakage, Inflammation of the gingiva adjacent to/around the space maintainer, Plaque accumulation around the band) will be taken into consideration. In order to evaluate the effects on periodontal tissues, pocket depth, plaque index values, gingival index values will be recorded and PLAP-1 and TNF-a levels in the gingival groove fluid will be examined for more detailed periodontal examination.

The total planned follow-up period is 18 months, with patients invited for follow-up appointments at six-month intervals.

Evaluations will be made at the end of the study with repeated measurements at baseline and control sessions.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy children
* Bilateral early loss of deciduous first molar teeth in the lower jaw
* Presence of radiographically confirmed permanent tooth germ under the extracted deciduous tooth
* Radiographically determined 1,5 mm minimum of bone existence above the permanent tooth germ
* Existence of flush terminal plane/mesial step in decidious dentition and Angle class 1 molar relationship in mixed dentition
* Existence of radiographically and clinically healthy abutment teeth
* Frankl score 3 and 4 children

Exclusion Criteria:

* Patients with systemic diseases
* Frankl score 1 and 2 children

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Clinical success | Up to 18 months
  The clinical success rate of appliances in terms of survival time by checking both space maintainers for these failure criteria: Dissolution of the bonding cement, loop distortion/breakage, separation/breakage from solder area ( for soldered conventional band and loop space maintainer).
Evaluation of periodontal tissue changes around both space maintainers according to the periodontal pocket depth measuring | Up to 18 months
  The pocket depth will be measured by probing the six sides of the teeth (mesio-buccal, mesio-lingual, disto-buccal, disto-lingual, mid-buccal, mid-lingual).
Evaluation of periodontal tissue changes around both space maintainers according to Plaque index values | Up to 18 months
  Plaque index, that is running in a scale from 0 to 3 where 0 means no plaque,1 film of plaque adhering to free gingival margin,2 moderate accumulation of soft deposits on the tooth and gingival margin, and 3 means abundance of soft debris.
Evaluation of periodontal tissue changes around both space maintainers according to the gingival index values | Up to 18 months
  In order to evaluate the effects of both space maintainers on periodontal tissues, gingival index values will be recorded at baseline, 6th, 12th and 18th months.
  Gingival index, scores from 0 to 3 where 0 no inflammation, 1slight redness no bleeding on probing, 2 redness and bleeding on probing, and 3 severe inflammation with edema and ulceration to spontaneous bleeding.
Evaluation of periodontal tissue changes around both space maintainers with gingival groove fluid examination | Baseline and 6.month
  For detailed periodontal evaluation, PLAP-1 and TNF-a levels in the gingival groove fluid will be examined at the baseline and 6th month visits. Gingival groove fluid samples will be taken from two separate points of the teeth which the bands of the band and loop space maintainers' had been placed, with PerioPaper strips. Afterwards, the strips taken from each tooth will be packaged separately in eppendorf tubes and stored at -80 degrees until it is time to evaluate. The samples will be evaluated by ELISA tests then the results will be compared.

SECONDARY OUTCOMES:
Measuring space maintaining efficiency | Up to18 months
  With the help of a digital caliper, the contact points of the teeth adjacent to the extraction space will be measured and the effective protection of the space will be monitored. First measurement will be done right before the space maintainers' placement. The caliper measurement will be repeated at the 6th, 12th and 18th months.
Comparing the two impression methods in terms of patient satisfaction. | Immediately after the impression procedure
  Two different impression methods will be used for the two techniques in the impression phase required for the production of the space maintainers. For the appliance to be produced with a three-dimensional printer, digital impressions will be taken with 3Shape intraoral scanner. For the conventional space maintainer production, impressions will be taken with traditional impression spoons using alginate material. With the help of a Likert scale from 1 to 5(with the help of smiley faces), the satisfaction levels of the children about the impression phases will be measured right after the impression process finished.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Aydin, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No